CLINICAL TRIAL: NCT05009836
Title: A Multicenter, Randomized, Double-blind, Phase III Clinical Study to Evaluate the Efficacy and Safety of Savolitinib + Osimertinib Versus Placebo + Osimertinib as the First Line Therapy for Patients With EGFRm+/MET+ NSCLC
Brief Title: Clinical Study on Savolitinib + Osimertinib in Treatment of EGFRm+/MET+ Locally Advanced or Metastatic NSCLC
Acronym: SANOVO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-504-00CH4
Record Dates: First submitted 2021-07-30; First posted 2021-08-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 320 patients, and eligible patients will be randomized in a ratio of 1:1 into the following treatment groups using central randomization system (IWRS): • Study group: Savolitinib 600 mg or 400 mg QD orally + Osimertinib 80 mg QD orally
  • Control group: placebo 600 mg or 400 mg QD orally + Osimertinib 80 mg QD orally
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Savolitinib (Experimental): Savolitinib 600 mg or 400 mg QD orally +Osimertinib 80 mg QD orally ( every 3 weeks)
  Interventions: Drug: Savolitinib
- placebo (Placebo Comparator): placebo 600 mg or 400 mg QD orally+ Osimertinib 80 mg QD orally ( every 3 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Savolitinib — Subjects will receive Savolitinib orally once per day (QD) + Osimertinib orally QD,21day cycles (every 3 weeks) until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Other Names: HMPL-504
  Arms: Savolitinib
Drug: Placebo — Subjects will receive placebo orally once per day (QD) + Osimertinib orally QD,21day cycles (every 3 weeks) until disease progression, death, adverse
  Arms: placebo

SUMMARY:
A Phase III Clinical Study on Savolitinib Combined with Osimertinib in Treatment of EGFRm+/MET+ Locally Advanced or Metastatic Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Phase III Clinical Study to Evaluate the Efficacy and Safety of Savolitinib Combined with Osimertinib versus Placebo Combined with Osimertinib as the First-line Therapy for Patients with EGFRm+/MET+ Locally Advanced or Metastatic Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware of this study and voluntary to sign the informed consent form, and being willing and able to comply with the study procedure;
2. Age ≥ 18
3. In accordance with the Eighth Edition of TNM Staging of Lung Cancer by the International Association for the Study of Lung Cancer and American Joint Committee on Cancer, and patients with histologically or cytologically confirmed unresectable locally advanced (stage ⅢB/ⅢC), metastatic or recurrent (stage IV) NSCLC who are not suitable for radical concurrent chemoradiotherapy;
4. Carrying two common EGFR mutations clearly related with the sensitivity to EGFR-TKI (i.e., exon 19 deletion, and L858R) and c-MET overexpression
5. Having measurable lesions (in accordance with RECIST 1.1 criteria);
6. ECOG Performance Status score 0 or 1, or Karnofsky score ≥80;
7. Survival is expected to exceed 12 weeks;
8. No any previous systematic antitumor therapy for advanced/metastatic disease;
9. adequate bone marrow reserve or organ function
10. Female patients of childbearing potential must agree to use effective contraceptive methods from screening period to 4 weeks after discontinuation of the study drug 11. Male patients whose sexual partners are women of childbearing potential must use condoms during sexual intercourse during the study and within 6 months after discontinuation of study drug

12. Being able to take or swallow the drug orally.

Exclusion Criteria:

1. Previous treatment with EGFR inhibitors or MET inhibitors;
2. Currently having other malignant tumors, or having other infiltrating malignant tumors in the past 5 years
3. Antitumor therapy within 2 weeks prior to the start of study treatment, including hormone therapy, biotherapy, immunotherapy or the traditional Chinese medicine for antitumor indication;
4. Having received extensive radiotherapy (including radionuclide therapy, e.g., Sr-89) within 4 weeks prior to the start of study treatment or palliative local radiotherapy within one week prior to the start of study treatment, or the above adverse reactions of radiotherapy did not recover;
5. Having received a major surgery within 4 weeks prior to the start of study treatment or a minor surgery (except biopsy, and venous catheterization) within one week prior to the start of study treatment;
6. Currently receiving the potent CYP3A4 inducers or potent CYP1A2 inhibitors within two weeks prior to the start of study treatment;
7. Having not been sufficiently recovered from the toxicity and/or complication resulting from any interventional measure prior to the start of treatment;
8. Clinically significant active infection, including but not limited to tuberculosis, human immunodeficiency virus (HIV) infection (positive HIV1/2 antibody);
9. Active hepatitis B, or active hepatitis C;
10. Acute myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack;
11. Uncontrollable hypertension despite the use of drugs,
12. Mean resting corrected QT interval (QTcF) or Any important abnormality in rhythm;
13. Patients whose known cancerous thrombus or deep vein thrombosis are stable for ≥2 weeks after receiving treatment with low molecular weight heparin (LMWH) or analogues with similar efficacy can be enrolled;
14. Any important abnormality in rhythm
15. Presence of meningeal metastasis, spinal cord compression or active brain metastasis prior to the start of study treatment.
16. Known allergy to the active or inactive ingredient of Savolitinib or Osimertinib;
17. Lack of compliance with participation in this clinical study or inability to comply with the limitations and requirements of the study, as judged by investigators;
18. Having participated in other drug clinical trials and received the study drug within 3 weeks prior to the start of study treatment; 19. Known allergy to the active or inactive ingredient of Savolitinib or Osimertinib; 20. Previous history of interstitial lung diseases, drug-induced interstitial lung diseases, radiation pneumonitis requiring glucocorticoid therapy and any active interstitial lung diseases; 21. Pregnant and lactating women; 22. Any other disease, metabolic abnormality, physical examination abnormality or laboratory examination abnormality, certain disease or state, based on which there is a reason to suspect that the subject is not suitable for the study drug, or one condition that will affect intepretaton of the study results or put the subject at high risk.

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 320 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 17 months after the last patient enrolled
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Safety and tolerability | 17 months after the last patient enrolled
  Incidence and nature of treatment emergent adverse events (TEAE), the other safety variables including physical examination, vital signs and laboratory examinations
The objective response rate of the tumor (ORR) | 17 months after the last patient enrolled
  the incidence of confirmed complete response or partial response
The disease control rate (DCR) | 17 months after the last patient enrolled
  the incidence of complete response, partial response and stable disease
Duration of Response (DoR) | 17 months after the last patient enrolled
  the duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded
Overall survival (OS) | 17 months after the last patient enrolled
  the time from the date of randomization to the date of death (all causes)
Time to Response (TTR) | 17 months after the last patient enrolled
  the period from the date of randomization to the date when the criteria for complete response or partial response was first measured (first record shall prevail).
PFS | 17 months after the last patient enrolled
  Progression-free survival (PFS) using IRC as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Development of diagnostic technology | 17 months after the last patient enrolled
  The residual samples may be used for development of MET Companion Diagnostics (CDx)

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No